CLINICAL TRIAL: NCT03027466
Title: Integrating Use of Self-Affirmation Content Into a Mobile App to Promote Quit Attempts With Text-Based Smoking Cessation Intervention Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Klein, Ph.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 999917039; 17-C-N039
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Results first posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Number of Quit Attempts
Keywords: Quitting Smoking; Phone Application
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baseline Affirmation and Affirmation Texts (Experimental): Participants will be given a "Baseline Affirmation" Quiz at the beginning of the study and will receive affirmation text messages throughout the study
  Interventions: Behavioral: Self-affirmation induction
- Baseline Affirmation and No Affirmation Texts (Active Comparator): Participants will be given a "Baseline Affirmation" Quiz at the beginning of the study but will not receive affirmation text messages throughout the study
  Interventions: Behavioral: Self-affirmation induction
- No Baseline Affirmation and Affirmation Texts (Active Comparator): Participants will not be given a "Baseline Affirmation Quiz" but will receive affirmation text messages throughout the study
  Interventions: Behavioral: Self-affirmation induction
- No Baseline Affirmation and No Affirmation Texts (Placebo Comparator): Participants will experience the Smoke Free United Kingdom (UK) app without any affirmation content Smoke Free UK app (no baseline affirmation quiz and no affirmation text messages)
  Interventions: Behavioral: Self-affirmation induction

INTERVENTIONS:
Behavioral: Self-affirmation induction — Participants will be randomly assigned to one of 4 conditions as part of a 2 (Integrated affirmation: Affirmation texts present versus absent) X 2 (Baseline affirmation: questionnaire present versus absent) design (these affirmations are described below). Those in the control condition will receive no changes to the app (standard of care control condition). Booster affirmation: Participants will receive an integrated affirmation every time they spontaneously report experiencing a craving. These will show up in a screen that shows Tips. We will be able to assess how many times participants reported experiencing a craving and thus saw a booster message.

SUMMARY:
Background:

Quitting smoking is hard. It is easy to relapse. Smokers may think of temptation to smoke as a threat if they think it suggests that they are unable to meet the challenges of stopping. When people feel such a threat to their sense of self-identity, they may get defensive. They may want to downplay the importance of quitting. This could make them try to quit less. Self-affirmation is a process of focusing on strengths and values. This can offset threats to the self and promote healthier behavior.

Objective:

To explore people s values, smoking attitudes, and smoking behavior.

Eligibility:

People ages 18 and older who smoke

Design:

The study takes place entirely on a mobile device.

Participants will give their age, gender, data about their smoking habits, and desired quit date.

Then they will get different texts about quitting.

Participants will answer follow-up surveys 1 and 3 months later.

...

DETAILED DESCRIPTION:
Quitting smoking is challenging and relapse is likely. Smokers may perceive temptation to smoke as threatening if they think it suggests that they are unable to meet the challenges of cessation. When individuals experience such a threat to their sense of self-identity (e.g., to their sense that they have integrity and/ or competence), they often respond defensively. Individuals have a tendency to react defensively to information that informs them that their behavior increases risk for a particular disease or negative health consequences. Self-affirmation a process through which individuals focus on their strengths and values can offset threats to the self and promote healthier behaviors, including smoking cessation. To the extent that relapse or difficulty quitting is perceived as a threat to self-identity, when individuals are presented with the opportunity to self-affirm they may perceive failure as less threatening, mitigating the motivation to downplay the importance of quitting. Preliminary evidence suggests that self-affirmation can be feasibly incorporated into an existing smoking cessation text message-based intervention, and may bolster cessation rates among users motivated to quit smoking. Here, we propose to extend that research by examining whether the addition of self-affirmation text messages to a smoking cessation app (Smoke Free United Kingdom (UK) promotes smoking cessation, compared to standard of care (i.e., existing app content only). Importantly, self-affirmation material will be incorporated into the current app and will not change the goals or nature of the original texting program. We predict that the individuals in the self-affirmation condition will be more likely to report being smoke-free at the 1-month and 3-month follow-ups.

ELIGIBILITY:
* INCLUSION/EXCLUSION:
* Because the app is designed to assist with smoking cessation, all smokers are eligible to participate.
* Subjects are eligible if they are 18+ years of age.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7899 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M Klein, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armitage CJ, Harris PR, Hepton G, Napper L. Self-affirmation increases acceptance of health-risk information among UK adult smokers with low socioeconomic status. Psychol Addict Behav. 2008 Mar;22(1):88-95. doi: 10.1037/0893-164X.22.1.88. PMID 18298234
- [Background] Spohr SA, Nandy R, Gandhiraj D, Vemulapalli A, Anne S, Walters ST. Efficacy of SMS Text Message Interventions for Smoking Cessation: A Meta-Analysis. J Subst Abuse Treat. 2015 Sep;56:1-10. doi: 10.1016/j.jsat.2015.01.011. Epub 2015 Feb 2. PMID 25720333
- [Background] Cohen GL, Garcia J, Purdie-Vaughns V, Apfel N, Brzustoski P. Recursive processes in self-affirmation: intervening to close the minority achievement gap. Science. 2009 Apr 17;324(5925):400-3. doi: 10.1126/science.1170769. PMID 19372432
- [Result] Seaman EL, Robinson CD, Crane D, Taber JM, Ferrer RA, Harris PR, Klein WMP. Association of Spontaneous and Induced Self-Affirmation With Smoking Cessation in Users of a Mobile App: Randomized Controlled Trial. J Med Internet Res. 2021 Mar 5;23(3):e18433. doi: 10.2196/18433. PMID 33666561

RESULTS

PARTICIPANT FLOW:
Groups:
- Baseline Affirmation and Affirmation Texts: Participants will be given a "Baseline Affirmation" Quiz at the beginning of the study and will receive affirmation text messages throughout the study
  Self-affirmation induction: Participants will be randomly assigned to one of 4 conditions as part of a 2 (Integrated affirmation: Affirmation texts present versus absent) X 2 (Baseline affirmation: questionnaire present versus absent) design (these affirmations are described below). Those in the control condition will receive no changes to the app (standard of care control condition).Booster affirmation: Participants will receive an integrated affirmation every time they spontaneously report experiencing a craving. These will show up in a screen that shows Tips. We will be able to assess how many times participants reported experiencing a craving and thus saw a booster message.
Period: Overall Study
Arm/Group | Baseline Affirmation and Affirmation Texts | Baseline Affirmation and No Affirmation Texts | No Baseline Affirmation and Affirmation Texts | No Baseline Affirmation and No Affirmation Texts
Started | 2027 | 1984 | 1903 | 1985
Completed | 158 | 165 | 160 | 164
Not Completed | 1869 | 1819 | 1743 | 1821
Not completed — Opting out of the app | 1869 | 1819 | 1743 | 1821

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline Affirmation and Affirmation Texts | Baseline Affirmation and No Affirmation Texts | No Baseline Affirmation and Affirmation Texts | No Baseline Affirmation and No Affirmation Texts | Total
Number analyzed (Participants) | 2027 | 1984 | 1903 | 1985 | 7899
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2027 | 1984 | 1903 | 1985 | 7899
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (8.6) | 30.5 (8.6) | 30.5 (8.8) | 30.5 (8.7) | 30.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 799 | 759 | 765 | 786 | 3109
  Male | 1228 | 1225 | 1138 | 1199 | 4790
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2027 | 1984 | 1903 | 1985 | 7899
Number of Participants Currently Using Cessation Aid [Count of Participants; unit: Participants]
  Yes | 446 | 401 | 434 | 440 | 1721
  No | 1581 | 1583 | 1469 | 1545 | 6178
Desire to Smoke [Mean (Standard Deviation); unit: units on a scale] — Desire to smoke: 1 = not at all; 5 = a lot.
  units on a scale | 3.2 (1.3) | 3.1 (1.4) | 3.2 (1.3) | 3.1 (1.4) | 3.2 (1.3)
Quit Attempts in Past Year [Mean (Standard Deviation); unit: Attempts] — Past year cessation attempts were assessed as a write-in question; all values from 0 to 365 were considered valid cases. All responses outside of this range were excluded from analysis of past year cessation attempts but were included in all subsequent analyses.
  Attempts | 7.2 (22.8) | 6.5 (20.7) | 6.6 (19.6) | 7.9 (27.5) | 7.9 (27.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting a Quit Attempt Within the Past Week at 1 Month and 3 Months
Description: Participants were asked to report the number of times they attempted to quit smoking at 1 month and 3 months.
Time Frame: 1 month and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Affirmation and Affirmation Texts | Baseline Affirmation and No Affirmation Texts | No Baseline Affirmation and Affirmation Texts | No Baseline Affirmation and No Affirmation Texts
Number analyzed (Participants) | 2027 | 1984 | 1903 | 1985
Participants
  Past Week Cessation at 1 Month | 142 | 143 | 139 | 145
  Past Month Cessation at 1 Month | 114 | 128 | 128 | 133
  Past Week Cessation at 3 Months | 54 | 58 | 55 | 48
  Past Month Cessation at 3 Months | 46 | 49 | 48 | 38

2. Secondary Outcome: Number of Days Participants Remained Smoke-free at the 1 and 3 Month Follow-up
Description: Participants were asked the number of days they have remained smoke-free at the 1 and 3 month follow-up.
Time Frame: 1 month and 3 months follow-up
Population: This outcome measure was not done because there was too little variability, and the data could not be analyzed due to high levels of attrition. The former Principal Investigator left the institute and no data are available or will ever become available for this Outcome.
Arm/Group | Baseline Affirmation and Affirmation Texts | Baseline Affirmation and No Affirmation Texts | No Baseline Affirmation and Affirmation Texts | No Baseline Affirmation and No Affirmation Texts
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Type of Tobacco Products
Description: Participants will be asked the type of tobacco products they use at the 1 and 3 month follow-up.
Time Frame: 1 month and 3 months follow-up
Population: This outcome measure was not done because type of tobacco products were not collected from participants at 1 month and 3 months follow-up.
Arm/Group | Baseline Affirmation and Affirmation Texts | Baseline Affirmation and No Affirmation Texts | No Baseline Affirmation and Affirmation Texts | No Baseline Affirmation and No Affirmation Texts
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Study start to study completion date, approximately 17 months and 26 days.
Arm/Group | Baseline Affirmation and Affirmation Texts | Baseline Affirmation and No Affirmation Texts | No Baseline Affirmation and Affirmation Texts | No Baseline Affirmation and No Affirmation Texts
All-Cause Mortality (participants affected / at risk) | 0/2027 | 0/1984 | 0/1903 | 0/1985
Serious Adverse Events (participants affected / at risk) | 0/2027 | 0/1984 | 0/1903 | 0/1985
Other Adverse Events (participants affected / at risk) | 0/2027 | 0/1984 | 0/1903 | 0/1985

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT03027466/Prot_SAP_000.pdf